CLINICAL TRIAL: NCT05291585
Title: Safety and Efficacy of the Dedicated Venous Sinus Thrombectomy Stent for Endovascular Treatment of Cerebral Venous Sinus Thrombosis.
Brief Title: The Dedicated Venous Sinus Thrombectomy Stent for Endovascular Treatment of Cerebral Venous Sinus Thrombosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVST-EVT
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Venous Sinus Thrombosis
Keywords: cerebral venous sinus thrombosis; endovascular treatment; thrombectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the dedicated venous sinus thrombectomy stent (Experimental): Patients diagnosed with acute or subacute venous sinus thrombosis within 28days from the onset of symptoms to endovascular treatment, regardless of whether anticoagulation has been performed. The dedicated venous sinus thrombectomy stent can be used to remove the thrombus to restore sinus blood flow.
  Interventions: Device: the dedicated venous sinus thrombectomy stent
- balloon catheter thrombectomy (Active Comparator): Intracranial thrombectomy was balloon catheter in conjunction with aspiration performed with a control product
  Interventions: Device: balloon catheter thrombectomy

INTERVENTIONS:
Device: the dedicated venous sinus thrombectomy stent — the dedicated venous sinus thrombectomy stent in conjunction with aspiration for CVST patients within 28 days of symptom onset.
  Arms: the dedicated venous sinus thrombectomy stent
Device: balloon catheter thrombectomy — Intracranial thrombectomy was conducted by using a balloon catheter in conjunction with aspiration as control group.
  Arms: balloon catheter thrombectomy

SUMMARY:
A prospective, single-center, open-label,randomized, controlled,non-inferiority clinical trial will be conducted to evaluate the safety and efficacy of a dedicated venous sinus thrombectomy stent for endovascular treatment of cerebral venous sinus thrombosis.

DETAILED DESCRIPTION:
Endovascular mechanical thrombectomy is reserved for the treatment of refractory cerebral venous sinus thrombosis (CVST) in the scenario of clinical deterioration in spite of appropriate anticoagulant therapy. However, due to the vascular anatomic and pathophysiological differences, the present used devices,such as stent retriever for arterial occlusion ,aspiration system and balloon catheter cannot provide optimal restoration of venous outflow for high load venous sinus thrombosis.This is a prospective, single-center, open-label, randomized, controlled , non-inferiority clinical trial to evaluate the safety and efficacy of the dedicated venous sinus thrombectomy stent ,which is a novel NiTi- braided Stent Retriever compared to balloon catheter used before in our center. Patients are eligible if they have a radiologically proven CVST, a high probability of poor outcome.

The trial aims to randomize 60 patients with a 1:1 allocation to receive the dedicated venous sinus thrombectomy stent or balloon catheter.

The primary outcome is the success rate of immediate recanalization.The most important secondary outcomes are mRS and mortality rate at 90 days. The intracranial hemorrhage and other adverse events after post-operative 24 hours and 7 days are the principal safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral venous sinus thrombosis (from onset to randomization less than 28 days) confirmed by cerebral angiography, magnetic resonance venography or computed tomographic venography
2. Severe form of CVT with a high chance of incomplete recovery, as defined by the presence of one or more of the following risk factors

   1. Clinical deterioration or progression despite anticoagulation
   2. Stupor, Coma (Glasgow coma scale < 9) or mental status disorder
   3. Involvement of multiple sinus veins results in severe high cranial pressure and rapid vision loss
   4. Venous infarction or intracranial hemorrhage with high load venous sinus thrombosis
   5. Thrombosis of the straight sinus
3. The subject (or his/her guardian) agrees to participate in this study and signs the informed consent

Exclusion Criteria:

Age less than 18 years Duration from onset to randomization more than 28 days Recurrent CVST Pregnancy (women in the puerperium may be included) Isolated cavernous sinus thrombosis or isolated cortical vein thrombosis Clinical and radiological signs of impending transtentorial herniation due to large space-occupying lesions and 4th ventricle compression and hydrocephalus, which requires emergency surgery Recent (< 2 weeks) major surgical procedure (does not include lumbar puncture) or severe cranial trauma Contraindication for anti-coagulant or thrombolytic treatment

1. documented generalized bleeding disorder
2. concurrent thrombocytopenia (<100 x 10E9/L)
3. severe hepatic or renal dysfunction, that interferes with normal coagulation
4. gastrointestinal tract hemorrhage (< 3 months, not including hemorrhage from rectal hemorrhoids) Any known serious condition (such as terminal cancer) with a poor short term (1 year) prognosis independent Known allergy against contrast used during endovascular procedures or the thrombolytic or anticoagulation drug used Previously legally incompetent prior to CVST No informed consent Other conditions judged by the researcher to be unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Success rate of immediate recanalization | immediately intra-operative
  3-grade classification scheme that considers different grades for patients with complete recanalization, partial recanalization and no recanalization.
  Complete recanalization defined as blood flow without any interruption, Partial recanalization defined as small interruptions of continuous blood flow and narrowing of the venous lumen No recanalization defined as interrupted blood flow.

SECONDARY OUTCOMES:
The proportion of functional independence (modified Rankin score 0-2) | up to 7 days and 90 days post-procedure
  0-No symptoms; 1-No significant disability; 2-Slight disability; 3-Moderate disability; 4-Moderately severe disability; 5-Severe disability; 6-Dead.
The time of thrombectomy procedure | intra-operative
  The time of thrombectomy procedure refers to the time from entry of thrombectomy device to vascular recanalization) or the end time of surgery for patients with no vascular recanalization
Changes in NIHSS score | pre-procedure, up to 7 days and 90 days post-procedure
  Changes in NIHSS score 7days or at discharge and 90 days post-procedure compared with pre-procedure.
Success rate of instrument operation | intra-operative
  Device operation success = the number of devices completed conveying to the occlusive segment of the sinus, releasing and retracting in the group/the number of all test devices used in the group ×100%
The proportion of symptom-free and improved | up to 7 days and 90 days post-procedure
  The symptoms include headache, visual dysfunction, tinnitus, cognitive disorder and epilepsy, etc.
CSF opening pressure | up to 7days
  Change of CSF opening pressure 7 days or at discharge post-procedure compared with pre-procedure by lumbar puncture
Modified Rankin Scale | up to 7 days and 90 days post-procedure
  Distribution of Modified Rankin Scale
The incidence of symptomatic intracranial hemorrhage | within 7 days post-procedure
  Symptomatic intracranial hemorrhage within 7 days post-procedure, specifically intracranial hemorrhage (intracranial parenchymal hematoma, subarachnoid hemorrhage, an ventricular hemorrhage) accompanied by neurological deterioration (NIHSS score increased by ≥4 points compared with pre-procedure.
Peri-procedural complications | intra-operative and 7 days post-procedure
  Procedure associated complications: vasospasm, dissection, perforation and emboli to new territory.
All cause mortality | within 90 days post-procedure
  All cause mortality within 90 days post-procedure
Incidence of device defects | intra-operative
  Defects of research devices during clinical trials, such as operational difficulties, broken devices and any incident related with device defects.
Incidence of SAE (serious adverse events) or AE (adverse events) | intra-operative, 24 hours, 7 days and 90 days post-procedure
  Incidence of SAE (serious adverse events) or AE (adverse events) intra-operative, 24 hours, 7 days and 90 days post-procedure
The recurrence rate of CVST | up to 7 days and 90 days post-procedure
  The recurrence rate of CVST confirmed by clinical manifestations and imaging examinations

OTHER OUTCOMES:
CVST pathological markers | pre-procedure, intra-operative, up to 7 days
  CVST pathological markers of blood, clot and cerebral spinal fluid(CRP,IL-6,NSE,NLR,etc.
Imaging database | pre-procedure and 90 days post-procedure
  neuroimaging: MRV/CTV

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ferro JM, Canhao P, Stam J, Bousser MG, Barinagarrementeria F; ISCVT Investigators. Prognosis of cerebral vein and dural sinus thrombosis: results of the International Study on Cerebral Vein and Dural Sinus Thrombosis (ISCVT). Stroke. 2004 Mar;35(3):664-70. doi: 10.1161/01.STR.0000117571.76197.26. Epub 2004 Feb 19. PMID 14976332
- [Background] Lee SK, Mokin M, Hetts SW, Fifi JT, Bousser MG, Fraser JF; Society of NeuroInterventional Surgery. Current endovascular strategies for cerebral venous thrombosis: report of the SNIS Standards and Guidelines Committee. J Neurointerv Surg. 2018 Aug;10(8):803-810. doi: 10.1136/neurintsurg-2018-013973. Epub 2018 Jun 5. No abstract available. PMID 29871990
- [Background] Coutinho JM, Zuurbier SM, Bousser MG, Ji X, Canhao P, Roos YB, Crassard I, Nunes AP, Uyttenboogaart M, Chen J, Emmer BJ, Roosendaal SD, Houdart E, Reekers JA, van den Berg R, de Haan RJ, Majoie CB, Ferro JM, Stam J; TO-ACT investigators. Effect of Endovascular Treatment With Medical Management vs Standard Care on Severe Cerebral Venous Thrombosis: The TO-ACT Randomized Clinical Trial. JAMA Neurol. 2020 Aug 1;77(8):966-973. doi: 10.1001/jamaneurol.2020.1022. PMID 32421159
- [Background] Fan Y, Yu J, Chen H, Zhang J, Duan J, Mo D, Zhu W, Wang B, Ouyang F, Chen Y, Lan L, Zeng J; Chinese Stroke Association Stroke Council CVST Guideline Writing Committee. Chinese Stroke Association guidelines for clinical management of cerebrovascular disorders: executive summary and 2019 update of clinical management of cerebral venous sinus thrombosis. Stroke Vasc Neurol. 2020 Jun;5(2):152-158. doi: 10.1136/svn-2020-000358. Epub 2020 May 13. PMID 32409571
- [Background] Goyal M, Fladt J, Coutinho JM, McDonough R, Ospel J. Endovascular treatment for cerebral venous thrombosis: current status, challenges, and opportunities. J Neurointerv Surg. 2022 Aug;14(8):788-793. doi: 10.1136/neurintsurg-2021-018101. Epub 2022 Jan 12. PMID 35022302
- [Derived] Xu Y, Wu Y, Jiang M, Song B, Li C, Wu C, Duan J, Meng R, Zhou C, Li S, Yan F, Chen J, Li M, Ji X. Efficacy and Safety of a Dedicated Device for Cerebral Venous Thrombectomy: A Pilot Randomized Clinical Trial. Stroke. 2025 Jan;56(1):5-13. doi: 10.1161/STROKEAHA.124.045607. Epub 2024 Nov 27. PMID 39601121